CLINICAL TRIAL: NCT01370187
Title: Montelukast for Acute Bronchiolitis and Postbronchiolitis Viral Induced Wheezing in Infants 3 to 12 Months of Age in Bandar Abbas Children' Hospital
Brief Title: Montelukast for Acute Bronchiolitis and Postbronchiolitis Viral Induced Wheezing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hormozgan University of Medical Sciences (Other)
Responsible Party: Ali Asghar Parhiz, Hormozgan University of Medical Sciences (HUMS)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Montelukast for bronchiolitis
Record Dates: First submitted 2011-06-06; First posted 2011-06-09 (Estimated); Last update posted 2011-06-14 (Estimated); Status verified 2010-06

CONDITIONS: Bronchiolitis; Wheezing; Cough
Keywords: Bronchiolitis; Postbronchiolitis wheezing; Montelukast
MeSH Terms: conditions — Bronchiolitis; Respiratory Sounds; Cough | interventions — montelukast

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Control group
- Montelukast (Experimental): 4mg Montelukast daily for 2 months
  Interventions: Drug: Montelukast

INTERVENTIONS:
Drug: Montelukast — Montelukast 4mg daily for 2 months
  Arms: Montelukast

SUMMARY:
The aim of the current study is to evaluate the effect of Montelukast in treatment of acute bronchiolitis and postbronchiolitis viral induced wheezing of infants 3 to 12 months of age in Bandar Abbas Children' hospital.

DETAILED DESCRIPTION:
All the patients will be evaluated at the baseline, during hospitalization (daily) and at 2 months and 6 months after starting the intervention.

ELIGIBILITY:
Inclusion Criteria:

* infant in 3-12 months of age with first episode of wheezing or bronchiolitis
* written informed consent by parents

Exclusion Criteria:

* Previous wheezing episode or confirmed asthma or bronchiolitis
* recent bronchodilator use
* immune deficient
* immunosuppressive drug use
* croup or pneumonia diagnosis
* loss of follow up

Ages: 3 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 146 (Actual)
Dates: Start 2010-07; Primary Completion 2011-04 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Respiratory Distress Severity Score (RDSS) | participants will be followed for the duration of hospital stay, an expected average of 3 days
  RDSS is measured by wheezing (0, 1, 2)+ Cough (0, 1, 2)+Retraction (0, 1,2)+Respiratory rate(0,1,2)+ Oxygen saturation(0,1,2) scores

SECONDARY OUTCOMES:
average number of cough daily= as expressed parents during visits | 6 months
  none= No cough, Mild=less than 10 daily, Severe=More than 10 daily
Wheezing severity in the physical examination by physician | 6 Months
  None= no wheezing, Mild= mild expiratory, Severe= inspiratory and expiratory

CONTACTS AND LOCATIONS:
Overall Officials: Ali Asghar Parhiz, Resident, Principal Investigator — Hormzgan University of Medical Sciences (HUMS)
Locations (1):
- Hormozgan University of Medical Sciences (HUMS), Bandar Abbas, Hormozgan, Iran